CLINICAL TRIAL: NCT01560884
Title: A Double Blind, Dose-Ranging, Phase 1 Study In Healthy Volunteers to Assess Safety and the Phosphate Binding Capacity of Lanthanum Dioxycarbonate (SPI-014, Renazorb)
Brief Title: Study to Assess the Safety and the Phosphate Binding Capacity of Renazorb
Acronym: SPI-014
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPI-RZB-11-101
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Safety; Phosphate Binding Capacity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group B (Active Comparator): Six subjects will be randomly assigned to receive SPI-014 3000 mg/day dose and 2 subjects to receive placebo
  Interventions: Drug: Renazorb 3000 mg/day
- Group C (Active Comparator): Six subjects will be randomly assigned to receive SPI-014 4500 mg/day dose and 2 subjects to receive placebo
  Interventions: Drug: Renazorb 4500 mg/day
- Group D (Active Comparator): Six subjects will be randomly assigned to receive SPI-014 6000 mg/day dose and 2 subjects to receive placebo
  Interventions: Drug: Renazorb 6000 mg/day
- Group A (Active Comparator): Six subjects will be randomly assigned to receive SPI-014 1500 mg/day dose and 2 subjects to receive placebo
  Interventions: Drug: Renazorb 1500 mg/day

INTERVENTIONS:
Drug: Renazorb 1500 mg/day — Six subjects will be randomly assigned to receive SPI-014 1500 mg/day dose and 2 subjects to receive placebo
  Other Names: Renazorb
  Arms: Group A
Drug: Renazorb 3000 mg/day — Six subjects will be randomly assigned to receive SPI-014 3000 mg/day dose and 2 subjects to receive placebo
  Other Names: Renazorb
  Arms: Group B
Drug: Renazorb 4500 mg/day — Six subjects will be randomly assigned to receive SPI-014 4500 mg/day dose and 2 subjects to receive placebo
  Other Names: Renazorb
  Arms: Group C
Drug: Renazorb 6000 mg/day — Six subjects will be randomly assigned to receive SPI-014 6000 mg/day dose and 2 subjects to receive placebo
  Other Names: Renazorb
  Arms: Group D

SUMMARY:
The purpose of this trial is to study safety, tolerability, and phosphate binding capacity of Renazorb (SPI-014) in healthy volunteers before conducting trials in patients with renal failure. Renal excretion of phosphate is expected to decrease and fecal excretion of phosphate is expected to increase after treatment.

DETAILED DESCRIPTION:
This is a double blind, dose-ranging study in healthy volunteers. Four sequential dose cohorts of 8 subjects each are planned. Six subjects will be randomly assigned to receive SPI-014 and 2 subjects to receive placebo within each cohort. The doses of SPI-014 will be 1500 mg/day (Group A), 3000 mg/day (Group B), 4500 mg/day (Group C) and 6000 mg/day (Group D), taken orally 3 times a day within 15 min after meals.

Following a screening period and evaluation of eligibility criteria, subjects will be admitted to the clinical research unit. From Day 1 to Day 10 subjects will be placed on a controlled phosphate diet (approved by a qualified dietician). From Day 1 to Day 5 (each day), 24 hour urine and feces will be collected at each voiding and pooled in separate containers for baseline phosphorus content. On Days 6 to 10, the subjects will receive SPI-014 or placebo within 15 minutes after each of the 3 main meals (see table below). From the morning of Day 8 to the morning of Day 13, 24 hour urine and feces will be collected for each day to determine phosphorus content. Subjects will be discharged on Day 13 and return 7 days later for an End-of-Study Visit on Day 20.

Starting dose will be 1500 mg/day. All safety data, including laboratory tests and adverse events, will be reviewed prior to escalation to the next cohort. After completion of first cohort, if no grades 3 AEs (vomiting and nausea) are observed in the first cohort on Day 20,Confidential 24 treatment of the second cohort begins. Similarly, third and fourth cohort will follow after the completion of the second and third cohort respectively.

Subjects will be admitted to the clinical research unit on Day -1 and remain at the clinical research unit until Day 13. From Day 1 to Day 10, subjects will consume a phosphate-controlled diet designed to provide 37.5 mmol (1200 mg) of elemental phosphorus per day (3 meals and 1 snack). The mean phosphorus contents of the meals are 12.1 mmol (387 mg), 8.6 mmol (275 mg), 12.0 mmol (416 mg), and 2.6 mmol (83 mg) for breakfast, lunch, dinner, and snack, respectively. With breakfast, the majority of the phosphorus is administered in milk. With the other meals phosphorus is primarily administered in solid food. During this 10-day treatment period subjects will be required to ingest all meals in their entirety.

The primary endpoint is phosphate binding capacity of SPI-014 as judged by levels of phosphorus in feces and urine. Phosphate excretion in urine is expected to go down and fecal excretion is expected to go up after treatment with SPI-014. Safety assessments are periodic physical examinations with vital sign measurements, safety laboratory tests, ECGs, AEs, and serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers ≥ 18 years of age without history of significant medical disease will be enrolled.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Efficacy | 6 Months
  Efficacy will be evaluated by comparing difference in urine and fecal phosphorous excretion before and after treatment.

SECONDARY OUTCOMES:
Serum concentrations of lanthanum. | 30 Days
Safety | 6 Months
  Safety will be evaluated by physical examinations, vital sign measurements, safety laboratory tests, ECGs, AEs, and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, Principal Investigator — PAREXEL, Harbor Hospital Center, Baltimore, MD 21225
Locations (1):
- PAREXEL International - Baltimore Early Phase Clinical Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Pergola PE, Joy MS, Garsd A, Hasal SJ, Khare A, Reddy G, Gupta P, Finn WF. Safety and Phosphate-Binding Capacity of Oxylanthanum Carbonate in Healthy Volunteers. Clin Transl Sci. 2025 Jan;18(1):e70116. doi: 10.1111/cts.70116. PMID 39727283